CLINICAL TRIAL: NCT06813339
Title: A Double Blind, Placebo-controlled Study to Investigate the Safety, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of UDP-003 in Healthy Human Participants and Patients
Brief Title: Placebo-controlled Study of Single and Multiple Ascending Doses of UDP-003 in Healthy Human Participants and Patients
Acronym: CTx-001
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cyclarity Therapeutics, Inc. (Industry)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTx-001
Record Dates: First submitted 2025-01-13; First posted 2025-02-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerotic Cardiovascular Disease; Acute Coronary Syndromes
Keywords: Atherosclerosis; 7-ketocholesterol (7KC); Cyclodextrin; Plaque burden reduction; Healthy Participants; Acute coronary syndrome
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UDP-003 (Experimental): UDP-003 will be administered to the participants randomised to this arm. UDP-003 is a formulated as a sterile solution for injection, 300 mg/mL. Volume of administration is weight dependent and target doses are 1-25 mg/kg.
  Interventions: Drug: UDP-003
- Placebo (Placebo Comparator): Placebo will be administered to the participants randomised to this arm. Placebo formulated as sterile solution for injection. Volume injected will match the volumes of UDP-003 for each panel and each participant.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UDP-003 — The UDP-003 finished product is clear, colourless to yellow liquid that is intended to be a sterile solution for IV bolus push administration in sterile water at a concentration of 300 mg/mL.
  Arms: UDP-003
Other: Placebo — Placebo will be provided as a sterile clear, colourless solution formulated to match viscosity of the UDP-003 solution.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if UDP-003 is safe in healthy human participants and patients, assess the pharmacokinetics (PK)/pharmacodynamics (PD) of UDP-003 in healthy human participants and patients and its potential efficacy in patients.

Researchers will compare UDP-003 to a placebo in a blinded manner.

This first in human, randomised, double-blind, placebo-controlled, prospective, single-centre trial with a modular dose-finding design will be conducted in 3 parts:

* Part 1: 6 cohorts of 6 healthy participants receiving Single Ascending Doses (SADs),
* Part 2: 3 cohorts of 12 healthy participants receiving Multiple Ascending Doses (MADs) (6 doses over 16 days),
* Part 3: 1 cohort of 12 participants diagnosed with acute coronary syndrome (ACS; non-ST elevation myocardial infarction [NSTEMI] or unstable angina) at least 12 months post-event receiving multiple doses (6 administrations of the 25 mg/kg dose over 16 days).

The planned duration of the study for each participant will be:

* 4 weeks for SAD Participants (1-day treatment period, 4-week safety follow-up)
* 6 weeks for MAD Participants (16-day treatment period,4-week safety follow-up)
* 28 weeks for MD Patients (16-day treatment period, 6-month safety follow-up) Prior to participants being randomised to panels of increasing doses, all safety data will be reviewed for completed panels.

DETAILED DESCRIPTION:
This trial's objective will be to collect the preliminary clinical safety and clinical pharmacology data. The study objective in the patient cohort is obtaining preliminary information on the safety of UDP-003 in those carrying a detectable plaque burden and obtaining preliminary indication of efficacy in respect to reducing the plaque burden.

This first in human, randomised, double-blind, placebo-controlled, prospective, single-centre trial with a modular dose-finding design will be conducted in 3 parts:

* Part 1: 6 cohorts of 6 healthy participants receiving SADs,
* Part 2: 3 cohorts of 12 healthy participants receiving MADs (6 doses over 16 days),
* Part 3: 1 cohort of 12 participants diagnosed with acute coronary syndrome (ACS; non-ST elevation myocardial infarction [NSTEMI] or unstable angina) at least 12 months post-event receiving multiple doses (6 administrations of the 25 mg/kg dose over 16 days). The SAD part will include healthy participants randomised to either active or placebo with a 2:1 ratio (24 active, 12 placebo) and the MAD and MD Patient parts with a 3:1 ratio (36 active, 12 placebo).

Prior to participants being randomised to panels of increasing doses, all safety data will be reviewed for completed panels. Within each dose group in the SAD portion of the study, sentinel dosing will be implemented wherein 2 participants (1 active, 1 placebo) will be dosed at least 24 hours before the remaining participants in the cohort. Dosing in the MAD portion of the study will commence only after the Data Safety Monitoring Committee (DSMC) reviews the safety data from the 5th (20 mg/kg) SAD cohort.

Investigational Products A. UDP-003, formulated as a sterile solution for injection, 300 mg/mL. Volume of administration is weight dependent and target doses are 1-25 mg/kg.

B. Placebo formulated as sterile solution for injection. Volume injected will match the volumes of UDP-003 for each panel and each participant.

The investigational products will be administered as intravenous (IV) bolus push injection, in a blinded manner to sitting or supine participants. Doses lower than the highest dose will be diluted with vehicle (identical to placebo) to ensure the same dosing volume per body mass across placebo and active groups. No fasting is required.

In the MD panels, a single IV bolus push injection will be administered on Days 1, 4, 7,10, 13 and 16.

ELIGIBILITY:
Inclusion Criteria:

(Healthy Participants (SAD and MAD cohorts)):

* Healthy adult males and females, 18 to 55 years of age (inclusive) at the time of screening.
* Medically healthy with relevant renal parameters tests not exceeding 1.5 X the upper limits and no clinically significant screening results (e.g., laboratory profiles, medical history, vital signs, ECGs, physical examination) as deemed by the Principal Investigator; one retest is permitted at investigator discretion.

(Participants with ACS (MD Patient cohort):

* Adult males and females, 40 to 79 years of age (inclusive) at the time of screening, diagnosed with acute coronary syndrome (ACS), at least 12 months post event (NSTEMI or unstable angina).
* Medically stable with no clinically significant screening results (e.g., laboratory profiles including relevant renal parameters and liver function tests, medical history, vital signs, ECGs, physical examination) as deemed by the Principal Investigator.
* Participants on a stable regimen and dose of ACS treatment including statins, anticoagulants, blood thinners, anti-platelets or other standard of care for 3 months prior to screening and for whom no change in this treatment is planned during the participation in the study.

Exclusion Criteria:

(Healthy Participants (SAD and MAD cohorts)):

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease as deemed by the Principal Investigator.
* History of myocardial infarction (MI), transient ischemic attack (TIA), stroke, or familial history of coronary artery disease or first-degree heart attack below the age of 60.
* Any clinically significant ECG abnormality at Screening
* Diabetic participants

(Patients (MD cohort):

* Percutaneous coronary intervention or diagnostic angiogram planned after screening.
* Documented episode of post-MI pericarditis in the 3 months before enrollment.
* Ongoing heart failure as defined by Class IV New York Heart Association
* History or presence of significant pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* Ongoing infection or febrile illness.
* Ongoing atrial fibrillation or flutter.
* History of MI, TIA, or stroke diagnosed within the 12 months prior to screening.
* History of or planned coronary artery bypass grafting.
* Any cardiac intervention or cardiac hospitalization in the past 12 months
* Any clinically significant ECG abnormality at Screening.
* Participants with contraindications to CTA.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety outcome measures (Adverse Events) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  Occurrence of adverse events (AEs) of any type and severity
Safety outcome measures (Vital Signs: Systolic Blood Pressure) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  SBP will be measured in mmHg
Safety outcome measures (Vital Signs: Diastolic Blood Pressure) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  DBP will be measured in mmHg
Safety outcome measures (Vital signs: Heart Rate) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  Heart Rate will be measured in bpm
Safety outcome measures (Vital signs: Respiratory Rate) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  RR will be measured in rpm
Safety outcome measures (Vital signs: Temperature) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  Body temperature will be measured in Celsius (0C)
Safety outcome measures (Clinical Laboratory Parameters) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  For parameters outside of the reference range an assessment of the significance (clinically significant / non-clinically significant) will be provided and all data outside the reference range of the clinical laboratory will be listed for all study participants
Safety outcome measures (ECG QTCF Interval) | From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  The QTcF interval will be calculated using the formula QTcF = QT/√R-R interval in seconds
Safety outcome measures (Injection site reactions) | From first dose administration (Day 1) through From enrolment through 4 weeks for SAD Participants, 6 weeks for MAD Participants and 28 weeks for MD Patients
  Assessment for signs of phlebitis, extravasation, infection and pain before, during and after intravenous administration is vital to ensure the patency and viability of the vein. The reactions will be assessed using the current FDA Toxicity Grading Scale provides a measure for classifying injection site AEs by four grades [Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe) and Grade 4 (life threatening)].
Safety outcome measures (Audiometry: PTA) | From enrolment through 24 hours post dose for SAD Participants (Day 2), 24 hours post dose for MAD and MD Patients Participants (Day 17),
  Air/Bone Pure-tone audiometry (PTA) conduction testing will be done at 250, 500, 1000, 3000, 4000, 6000 and 8000Hz
Safety outcome measures (Audiometry: HFA) | From enrolment through 24 hours post dose for SAD Participants (Day 2), 24 hours post dose for MAD and MD Patients Participants (Day 17),
  Bone/Air High-frequency audiometry (HFA) conduction testing will be done at 9000, 10 000, 11200 and 12500Hz, Tympanometry, Self-evaluation questionnaires (tinnitus handicap inventory [THI] and dizziness handicap inventory [DHI])
Safety outcome measures (Audiometry: Self-evaluation questionnaire (THI)) | From enrolment through 24 hours post dose for SAD Participants (Day 2), 24 hours post dose for MAD and MD Patients Participants (Day 17),
  Self-evaluation questionnaire: using Tinnitus Handicap Inventory [THI] questionnaire
Safety outcome measures (Audiometry: Self-evaluation questionnaire (DHI)) | From enrolment through 24 hours post dose for SAD Participants (Day 2), 24 hours post dose for MAD and MD Patients Participants (Day 17),
  Self-evaluation questionnaire: using Dizziness Handicap Inventory [DHI] questionnaire

SECONDARY OUTCOMES:
Pharmacokinetics Outcome Measures (Cmax) | Day 1 for the SAD and Days 1 and 16 for the multiple dosing parts
  The maximum concentration achieved by UDP-003 in a specified compartment area of the body after the drug has been administered and before the administration of a second dose
Pharmacokinetics Outcome Measures (Tmax) | Day 1 for the SAD and Days 1 and 16 for the multiple dosing parts
  Time at which maximum concentration of UDP is reached
Pharmacokinetics Outcome Measures (half-life (t1/2)) | Day 1 for the SAD and Days 1 and 16 for the multiple dosing parts
  The estimate of the time it takes for the concentration or amount in the body of that drug to be reduced by exactly one-half (50%).
Pharmacokinetics Outcome Measures (AUC0-t and AUC0-inf) | Day 1 for the SAD and Days 1 and 16 for the multiple dosing parts
  Area under the concentration curve (AUC0-t and AUC0-inf) reflects the actual body exposure to drug after administration of a dose of the drug and is expressed in mg*h/L
Pharmacokinetics Outcome Measures (Total Plasma Clearance (CL)) | Day 1 for the SAD and Days 1 and 16 for the multiple dosing parts
  The volume of drug cleared from blood or plasma in unit time
Pharmacokinetics Outcome Measures (Volume of Distribution (Vd)) | Day 1 for the SAD and Days 1 and 16 for the multiple dosing parts
  The participant's drug's propensity to either remain in the plasma or redistribute to other tissue compartments

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia